CLINICAL TRIAL: NCT06950021
Title: Safety & Performance of CANOpus PINtuition Surgical Marker Navigation (CANOPIN)
Brief Title: Safety & Performance of CANOpus PINtuition Surgical Marker Navigation
Acronym: CANOPIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sirius Medical Systems B.V. (Industry)
Collaborators: Avania B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CANOPIN; NL-MF-000010932 (Other: CCMO)
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Surgery; Lymph Node Excision
Keywords: Breast conserving surgery; magnetic seed localization; pintuition; breast sparing surgery; surgical localization; surgical navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary breast lesion and/or axillary lymph node localisation prior to surgical excision (Experimental): Device: CANOPUS Magnetic Marker by Sirius Medical Systems B.V.
  Placement of experimental device in primary breast lesion and/or axillary lymph node indicated for surgical removal and requiring localisation
  Interventions: Device: Magnetic seed

INTERVENTIONS:
Device: Magnetic seed — All patients enrolled will receive a single Sirius Canopus Marker with two anchors added to it for improved tissue fixation. Implantation will be done by a radiologist before breast conserving surgery, usually scheduled within a few days after Canopus Marker implantation. The Canopus Marker is removed with the specimen during the surgery.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and performance of the Canopus Marker in adult breast cancer patients who are scheduled for breast-conserving surgery. The main questions it aims to answer are:

1. Can the Canopus Marker be safely and effectively used to mark tissue for surgical removal?
2. What is the satisfaction level of radiologists, surgeons, and patients with the use of the Canopus Marker?

Participants will:

* Have the Canopus Marker implanted into the tumor or nearby tissue using ultrasound guidance.
* Undergo surgery where the Canopus Marker will help guide the surgeon to the tumor, and the marker will be removed along with the tumor. This surgery is performed using an FDA cleared and CE-marked detection device (Sirius Pintuition Detector).
* Attend a follow-up visit two weeks after surgery to assess any adverse events and overall satisfaction.

DETAILED DESCRIPTION:
Breast cancer remains one of the most prevalent malignancies affecting women worldwide, necessitating a range of treatment modalities to manage and combat the disease effectively. These modalities include surgery, radiation therapy, chemotherapy, hormone therapy, and targeted therapy. Among these, breast-conserving surgery (BCS), also known as lumpectomy, has become a cornerstone of breast cancer treatment. BCS involves the removal of the cancerous tissue while preserving as much of the breast as possible. This approach aims to achieve oncologic safety comparable to mastectomy while offering psychological and cosmetic benefits. The success of BCS has been augmented by advancements in imaging techniques and surgical tools, facilitating precise tumour localization and excision.

Over the years, various localization technologies have been developed to enhance the precision of breast cancer surgeries. Traditional methods like wire localization have been widely used but are often associated with discomfort and logistical challenges. Advances in medical technology have led to non-wire localization methods such as radioactive seed localization (RSL) and radar systems. The commercially available Sirius Pintuition system, using magnetic seed localization, involves inserting a small magnetic marker into the tumour site, detectable with a magnetic probe during surgery. This system aims to offer advantages like improved subject comfort, precise localization, and ease of use for surgeons. The investigational Canopus Marker, building on Sirius Pintuition's success, aims to further improve the precision and effectiveness of breast-conserving surgeries. The Canopus Marker incorporates additional anchoring mechanisms designed to enhance its stability during breast-conserving surgeries. These enhancements aim to mitigate any potential risk of dislodgement, while maintaining the marker's detectability and ease of use for surgeons.

The present investigation is only evaluating if the additional anchors added to the Pintuition Marker, which is the Canopus Marker, is also safe and performing as intended. Therefore, the present investigation will be similar in design as the study that was conducted to obtain the Pintuition System's CE mark. That is, a single-arm, open-label study in one centre in The Netherlands. The sample size (n=35) is determined to demonstrate that the Canopus Marker does not perform worse than the Pintuition Marker and other similar marker-based localization devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent for the investigation
2. Subject is at least 18 years of age
3. Subject is diagnosed with a single, pathologically confirmed unifocal breast tumour (DCIS or invasive)
4. Tumour is ultrasound visible
5. Subject is indicated for primary breast conserving surgery and/or targeted axillary dissection
6. Subject is indicated for preoperative localization using a single marker in the primary breast lesion and/or a single marker in an axillary lymph node

Exclusion Criteria:

1. Subject is lactating or pregnant
2. Subject is expected to have surgery scheduled more than 6 weeks after implantation of the Canopus Marker.
3. Subject has an ICD or other active implant such as a pacemaker less than 5 cm away from the intended target location(s)
4. Subject has a proven infection or clinically significant hematoma at or close to the intended target location(s)
5. Subject is expected to require an MRI scan in the period between implantation and surgery
6. Known hypersensitivity to Titanium or Nickel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Performance: Retrieval Rate | From enrolment to the follow-up visit at 2 weeks after surgery (estimated 3-5 weeks)
  Proportion of procedures in which the Canopus marker is present on post-operative specimen X-ray and only the Pintuition Detector is used during surgery.
  Hypothesis: => 85%
Safety: Investigational Device-Related Serious Adverse Device Effects | From enrolment to the follow-up visit at 2 weeks after surgery (estimated 3-5 weeks)
  Proportion of patients who experienced an investigational device-related serious adverse device effect as assessed by MedDRA. Hypothesis: none.

SECONDARY OUTCOMES:
Radiologist's Satisfaction | Post-procedural (implantation)
  The secondary performance endpoints and hypotheses of this clinical investigation include: an overall radiologist satisfaction score of ≥7 measured on a 10-point Likert scale or comparable index
Surgeon Satisfaction | Post-procedural (surgery)
  The secondary performance endpoints and hypotheses of this clinical investigation include: an overall surgical satisfaction score of ≥7 measured on a 10-point Likert scale or comparable index
Subject Satisfaction | At post-operative check (2 weeks follow-up visit)
  The secondary performance endpoints and hypotheses of this clinical investigation include: an overall subject satisfaction score of ≥7 measured on a 10-point Likert scale or comparable index
Safety: Adverse Events | From enrolment to the follow-up visit at 2 weeks after surgery (estimated 3-5 weeks)
  Secondary safety endpoints include the reporting of the incidence, severity and causal relationship of adverse events (AEs), adverse device effects (ADEs), serious adverse events (SAEs), unanticipated serious adverse device events (USADEs) and device deficiencies (DDs) in accordance with ISO 14155:2020 definitions
Accuracy of Placement | Post-procedural (implantation)
  Average distance between Canopus Marker centre and tumour centre on the two post-placement mammographic images in mm
Operative Time | Post-procedural (surgery)
  Minutes from first incision until wound closure
Transcutaneous Detection Succesful | Periprocedural (surgery)
  Proportion of procedures in which a reliable signal of the Canopus Marker is detected on the intact skin using the Pintuition Detector
Marker Dislodgements | Post-procedural (surgery)
  Proportion of procedures in which the Marker dislodged during the surgical procedure.
Reoperation Rate | From enrolment to the follow-up visit at 2 weeks after surgery (estimated 3-5 weeks)
  Second, separate surgical procedure of same lesion or area indicated after multidisciplinary discussion

CONTACTS AND LOCATIONS:
Locations (1):
- Rode Kruis Ziekenhuis, Beverwijk, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided